CLINICAL TRIAL: NCT01958229
Title: A Multicenter Open-label, Observational Study of Telbivudine Treatment Outcome in Patients With Chronic B Virus Infection
Brief Title: Efficacy Study of Telbivudine in Chronic Hepatitis B Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200910027M
Record Dates: First submitted 2013-10-01; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Hepatitis B; Roadmap Concept in Chronic Hepatitis B Treatment; 24-week PCR Negativity of Telbivudine; PCR Negativity at 52 and 104 Week; HBeAg Seroconversion Rate at 52 and 104 Week
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 c.c whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CHB patients without cirrhosis

SUMMARY:
This study is designed to support the optimal use of telbivudine by providing data to refine our understanding of telbivudine efficacy and resistance in real life clinical setting in patients with chronic hepatitis B with defined baseline characteristics and 24-week PCR negativity.

DETAILED DESCRIPTION:
This study will be multicenter, open-label and observational data collection of patients on telbivudine who meet baseline characteristics defined as the majority of patients seen in the clinic setting. Data collection will take place after enrollment, at Week 12, 24, 52, 76 and 104 for efficacy assessments. In patients who discontinue observational drug earlier, clinical information would be kept following for assessment as well.

Study purpose:

This study is designed to evaluate the efficacy of telbivudine in real-life clinical settings with the use of the Roadmap Concept in chronic hepatitis B treatment.

Objectives:

Primary:

To observe telbivudine's 2-year efficacy in real-world clinical setting of achieving HBV-DNA < 60 IU/ml and HBeAg seroconversion rate in patients with defined baseline characteristics and 24-week treatment PCR negativity as previously reported in GLOBE study's sub-analysis.

Secondary:

1. To observe the treatment outcomes.
2. To validate the result of super-responder trial.
3. To validate the Roadmap Concept.

Population:

The study population will consist of a representative group of 500 chronic hepatitis B patients with detectable HBsAg for more than 6 months who need telbivudine therapy based on investigators' judgment in 16 medical centers located in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 65 years of age
* Documented chronic hepatitis B defined by ALL of following:

  1. Clinical history compatible with compensated chronic hepatitis B
  2. Detectable serum hepatitis B surface antigen (HBsAg)> 6 months and at the screening visit.

Exclusion Criteria:

* Pregnant or nursing
* co-infection with hepatitis C virus (HCV) or HIV
* Clinical or imaging diagnosis of cirrhosis
* Evidence of decreased renal function of creatinine >(=)2x ULN

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis B patients without cirrhosis
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
PCR negativity | week 52
HBeAg seroconversion rate | week 52
PCR negativity | week 104
HBeAg seroconversion rate | week 104

SECONDARY OUTCOMES:
Rate of ALT normalization | week 52
Genotypic resistance | week 52
Rate of ALT normalization | week 104
Genotypic resistance | week 104

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Horng Kao, Professor, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan